CLINICAL TRIAL: NCT05505006
Title: Management of Preoperative Anaemia in Surgical Oncology as a Tool to Reduce Blood Transfusion Need
Brief Title: Management of Preoperative Anaemia in Surgical Oncology
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Fabiana Busti, Clinical researcher, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-2016-02361206
Record Dates: First submitted 2022-08-11; First posted 2022-08-17 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Anemia; Tumor
Keywords: anemia; surgical oncology; transfusion; patient blood management
MeSH Terms: conditions — Anemia; Neoplasms | interventions — ferric carboxymaltose; Folic Acid; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: * Institution of an Anemia Clinic to identify all cancer patients with anemia before surgery
  * Treatment of treatable causes of anemia in all cancer patients within three weeks before surgery; in particular, iron deficiency (ID), folate deficiency and B12 deficiency
  * Collection of data concerning transfusions in the peri-operative period
  * Collection of peri-operative outcomes such as in-hospital mortality, myocardial infarction, ischemic stroke, acute renal failure, pneumonia, or sepsis, and Hb levels at discharge
  * Comparison of data relating to transfusions and outcomes with those obtained in a historical cohort of anemic patients eligible for oncological surgery for malignant tumors, matched by age, sex, and pathology enrolled in the three years 2017-2019
  * Evaluation of hepcidin levels in anemic cancer patients (explorative aim)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patients with anemia (i.e. Hb <12 g/dl if females, <13 g/dL if males) (Experimental): Cancer patients eligible for surgery with anemia will be managed as follows:
  * s-ferritin <100 mcg/l or s-ferritin <500 mcg/l + TSAT<20% = i.v. iron (ferric carboxymaltose, dosage according to body weight and Hb level)
  * folate < 5 ng/ml = folate 5 mg per day for 1 month
  * B12 < 200 pg/ml = B vitamin complex 1 tablet per day for 1 month
  Patients will receive combined treatment if they have multiple deficiencies simultaneously.
  Patients without correctable deficiencies will not receive any treatment.
  Interventions: Drug: Ferric Carboxymaltose Injection; Drug: Folic acid; Drug: B12

INTERVENTIONS:
Drug: Ferric Carboxymaltose Injection — Anemic patients with ID will receive i.v. iron. Dosage will be based on Hb level and patient body weight.
  Other Names: i.v. iron
Drug: Folic acid — Anemic patients with folate deficiency will receive folic acid 5 mg per day for 1 month
  Other Names: Folate
Drug: B12 — Anemic patients with B12 deficiency will receive B vitamin complex 1 tablet per day for 1 month
  Other Names: cobalamin

SUMMARY:
Preoperative anemia is detrimental in surgical patients, and its treatment with transfusions can further worsen outcomes, including increased hospital stay and mortality. Transfusions are also highly costly. In 2010, the World Health Organization endorsed the adoption of Patient Blood Management (PBM) programs, i.e., patient-centered multidisciplinary activities, including recognition and treatment of preoperative anemia. While the latter has been proved effective in reducing transfusions in setting like elective orthopedic surgery, widespread adoption is still lacking. Moreover, little is known about surgical oncology, a particular setting posing unique challenging. This change-promoting project attempts to fill this knowledge gap by establishing a multidisciplinary team aimed at optimal management of preoperative anemia in hepatobiliary/pancreas/gastrointestinal/renal surgical oncology. The primary endpoint is the reduction of transfusions, along with safer patient outcomes as compared to the historical series.

DETAILED DESCRIPTION:
BACKGROUND: Preoperative anemia is frequent in patients undergoing major surgery, varying from nearly 35% in elective orthopedic surgery (EOS) to >75% in colon cancer. Mounting data have shown that anemia is independently associated with an increased risk of morbidity and mortality in surgical patients. This is true even for mild-degree anemia, which is frequently overlooked. Of note, treatment of anemia with transfusions does not ameliorate the risk but instead appears to raise further perioperative morbidity, hospital length of stay, and mortality. Transfusions have adverse immunomodulatory effects that can increase infectious complications or cancer recurrence. Indeed, it is increasingly recognized that transfusions are one of the most costly and overused treatments in modern medicine. This has led to the implementation of Patient Blood Management (PBM) programs, i.e., patient-centered, multidisciplinary activities to promote safe and evidence-based use of transfusions. Recognition and treatment of preoperative anemia is a significant pillar of PBM, with proven efficacy in certain types of surgery, i.e., EOS. This has been facilitated by recent advances in the knowledge of the pathophysiology of iron, whose deficiency represents a common and treatable form of anemia in surgical patients. Nevertheless, evidence is scanty in surgical patients with malignancies, a particular subgroup that poses unique challenges.

Hypothesis and Significance: Recognition and treatment of preoperative anemia in surgical oncology through a well-organized, multidisciplinary Anemia Clinic should decrease blood transfusions, ultimately leading to better clinical outcomes and cost savings.

METHODOLOGIES and STATISTICAL ANALYSES: Evaluation and treatment of preoperative anemia will be performed as follows: we will perform a minimum panel of exams, i.e., complete blood count (CBC), creatinine, C-reactive protein, ferritin, transferrin saturation (TSAT), and circulating folate/B12 levels, to assess the presence of anemia, and to identify potentially correctable causes. On the same day on which the patient performs lab analyses in the morning, the surgeon will alert the Anemia Clinic with the patient's ID digital code. Case-manager MD at Anemia Clinic will evaluate lab results as soon they become available (expected time 3-4 hours after blood drawing) through the e-health system. Anemic patients will be invited to attend the Anemia Clinic the day after. They will be clinically evaluated, and treatment for anemia will be immediately prescribed/performed.

Core statistical analyses regarding transfusion use and patients' outcomes will be entrusted to external independent statisticians through subcontract. The diagnostic performance of hepcidin will be investigated through Area Under the Curve Receiving Operating Characteristic (AUC-ROC) and its prognostic implications by Kaplan-Meier curves.

The duration of the presented project is calculated as 36 months and will be divided into 3 different milestones as follows:

* M1: Study organization and coordination among the Units (study protocol preparation, procedures implementation for managing patient flow across units).
* M2: 24 months of Patient Enrolment (evaluation of preoperative hematological parameters and suitable treatment, surgery, postoperative evaluation) and ad interim follow-up evaluation after 1 month from the surgery.
* M3: statistical evaluation of results, publication preparation, and evaluation of the possible implementation of new improved internal guidelines for treating anemia in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent
* Eligibility to elective surgery for malignant oncological pathology.

  * Presence of pre-operative anemia (Hb <12 g/dL females, <13 g/dL males)
  * Age >=18 years

Exclusion Criteria:

* Patients with chronic anemia, regularly transfused
* Patients with Hemochromatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2024-08-13 (Estimated); Study Completion 2024-08-13 (Estimated)

PRIMARY OUTCOMES:
Change in transfusion number compared to a historical cohort of patients enrolled in the three-year period 2017-2019 | up to 4 weeks after surgery
  Evaluate whether implementing a program for early recognition and management of preoperative anemia leads to a reduction in blood transfusions in surgical oncology compared to historical cohort enrolled before the project
Change in short-term (30 days) patients' outcomes (perioperative complications including infections, cardiovascular events, and mortality) compared to a historical cohort of patients enrolled in the three years 2017-2019 | up to 4 weeks after surgery
  Evaluate whether implementing a program for early recognition and management of preoperative anemia leads to an improvement in some patient's clinical outcomes after surgery compared to the historical cohort enrolled before the project
Change in length of stay in hospital compared to a historical cohort of patients enrolled in the three-year period 2017-2019 | up to 4 weeks after surgery
  Evaluate whether implementing a program for early recognition and management of preoperative anemia leads to a shortening in the duration of hospitalization after surgery compared to the historical cohort enrolled before the project
Change in Hb levels (g/dl) at discharge compared to a historical cohort of patients enrolled in the three-year period 2017-2019 | up to 4 weeks after surgery
  Evaluate whether implementing a program for early recognition and management of preoperative anemia leads to an improvement in Hb levels at discharge compared to the historical cohort enrolled before the project

OTHER OUTCOMES:
To evaluate the role of hepcidin in the pathophysiology of cancer-related anemia, and its potential role as prognostic parameter and in predicting the response to iron therapy | at patient enrollment and at hospital admission
  hepcidin levels

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shander A, Knight K, Thurer R, Adamson J, Spence R. Prevalence and outcomes of anemia in surgery: a systematic review of the literature. Am J Med. 2004 Apr 5;116 Suppl 7A:58S-69S. doi: 10.1016/j.amjmed.2003.12.013. PMID 15050887
- [Background] Musallam KM, Tamim HM, Richards T, Spahn DR, Rosendaal FR, Habbal A, Khreiss M, Dahdaleh FS, Khavandi K, Sfeir PM, Soweid A, Hoballah JJ, Taher AT, Jamali FR. Preoperative anaemia and postoperative outcomes in non-cardiac surgery: a retrospective cohort study. Lancet. 2011 Oct 15;378(9800):1396-407. doi: 10.1016/S0140-6736(11)61381-0. Epub 2011 Oct 5. PMID 21982521
- [Background] Spahn DR. Patient Blood Management: Success and Potential in the Future. Ann Surg. 2016 Aug;264(2):212-3. doi: 10.1097/SLA.0000000000001787. No abstract available. PMID 27163953
- [Background] Ness PM, Frank SM. Enhancing patient blood management: a long-term FOCUS. Lancet. 2015 Mar 28;385(9974):1157-9. doi: 10.1016/S0140-6736(14)62344-8. Epub 2014 Dec 9. No abstract available. PMID 25499166
- [Background] Anthes E. Evidence-based medicine: Save blood, save lives. Nature. 2015 Apr 2;520(7545):24-6. doi: 10.1038/520024a. No abstract available. PMID 25832389
- [Background] Clevenger B, Mallett SV, Klein AA, Richards T. Patient blood management to reduce surgical risk. Br J Surg. 2015 Oct;102(11):1325-37; discussion 1324. doi: 10.1002/bjs.9898. Epub 2015 Aug 27. PMID 26313653
- [Background] Vaglio S, Prisco D, Biancofiore G, Rafanelli D, Antonioli P, Lisanti M, Andreani L, Basso L, Velati C, Grazzini G, Liumbruno GM. Recommendations for the implementation of a Patient Blood Management programme. Application to elective major orthopaedic surgery in adults. Blood Transfus. 2016 Jan;14(1):23-65. doi: 10.2450/2015.0172-15. Epub 2015 Dec 15. No abstract available. PMID 26710356
- [Background] Girelli D, Nemeth E, Swinkels DW. Hepcidin in the diagnosis of iron disorders. Blood. 2016 Jun 9;127(23):2809-13. doi: 10.1182/blood-2015-12-639112. Epub 2016 Apr 4. PMID 27044621
- [Background] Gross I, Trentino KM, Andreescu A, Pierson R, Maietta RA, Farmer S. Impact of a Patient Blood Management Program and an Outpatient Anemia Management Protocol on Red Cell Transfusions in Oncology Inpatients and Outpatients. Oncologist. 2016 Mar;21(3):327-32. doi: 10.1634/theoncologist.2015-0406. Epub 2016 Feb 10. PMID 26865590
- [Background] Froessler B, Palm P, Weber I, Hodyl NA, Singh R, Murphy EM. The Important Role for Intravenous Iron in Perioperative Patient Blood Management in Major Abdominal Surgery: A Randomized Controlled Trial. Ann Surg. 2016 Jul;264(1):41-6. doi: 10.1097/SLA.0000000000001646. PMID 26817624
- [Background] Calleja JL, Delgado S, del Val A, Hervas A, Larraona JL, Teran A, Cucala M, Mearin F; Colon Cancer Study Group. Ferric carboxymaltose reduces transfusions and hospital stay in patients with colon cancer and anemia. Int J Colorectal Dis. 2016 Mar;31(3):543-51. doi: 10.1007/s00384-015-2461-x. Epub 2015 Dec 22. PMID 26694926